CLINICAL TRIAL: NCT02195323
Title: Administration of Autologous Bone Marrow Mesenchymal Stem Cells (BM-MSCs) in Patients With Chronic Kidney Disease (CKD)
Brief Title: Autologous Bone Marrow Derived Mesenchymal Stromal Cells (BM-MSCs) in Patients With Chronic Kidney Disease (CKD)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Royan Institute (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Royan-Kidney-004
Record Dates: First submitted 2014-07-17; First posted 2014-07-21 (Estimated); Last update posted 2016-01-05 (Estimated); Status verified 2015-11

CONDITIONS: Chronic Kidney Disease
Keywords: autologous bone marrow mesenchymal stem cells chronic kidney disease
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Injections, Intravenous

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- MSC recipient (Experimental): The patients with CKD who underwent intravenous injection of MSC.
  Interventions: Biological: Intravenous injection

INTERVENTIONS:
Biological: Intravenous injection — Intravenous injection of bone marrow derived MSC in patients with CKD.
  Other Names: Intravenous transplantation

SUMMARY:
This study was designed to provide confirmation of safety of mesenchymal stem cells (MSCs) therapy in chronic kidney disease (CKD).

DETAILED DESCRIPTION:
We will assess the 18-month safety and potential efficacy of autologous MSCs as a therapy for CKD. A total of 10 patients with CKD IV injection of high doses 2×106/kg of autologous MSCs t, which will be derived from biopsies of their bone marrow. Assessments will be performed at 1, 3, 6, 12 and 18 months after cell injection. Changes in Glomerular Filtration Rate (GFR) were evaluated by scan isotope.

ELIGIBILITY:
Inclusion Criteria:

* Male and Female
* CKD symptoms
* CKD confirmed with serum and urine analysis and GFR 25-60 mL/min/1.73 m2
* Patient's age between 25 - 60 years
* Ability to understand and willingness to sign consent from

Exclusion Criteria:

* Pregnant or lactating
* Basis disease such as diabetes, malignancy and autoimmune
* Unable to follow post-operative exercise regimen or return for evaluations

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2014-04; Primary Completion 2015-12 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
mass formation | 6months
  Evaluation the probability of mass formation due to MSC transplantation 6 months after cell injection.
Creatinin | 1 month
  Evaluation the rise of creatinin 1 month after cell transplantation.

SECONDARY OUTCOMES:
GFR | 6months
  Evaluation the increase of GFR 6 months after cell transplantation with scan isotope .

CONTACTS AND LOCATIONS:
Overall Officials: Hamid Gourabi, PhD, Study Chair — Head of Royan Institute; Nasser Aghdami, MD,PhD, Study Director — Head of regenerative medicine department &cell therapy center of Royan Institute; Atieh Makhloogh, MD, Study Director — Mazandaran University of Medical Sciences, Mazandaran, Iran; Reza Moghadasali, PhD, Principal Investigator — Department of Regenerative Medicine And Royan Cell Therapy Center Royan Institute For stem Cell Biology and Technology
Locations (1):
- Royan Institute, Tehran, Iran

REFERENCES:
- See also: Related Info — http://Royaninstitute.org